CLINICAL TRIAL: NCT01253330
Title: Study of the Usage, Usability, Acceptability, and Effect on Adherence and Clinical Outcomes of a Web Based Text Messaging System for Adolescents With Asthma- Phase 2
Brief Title: Usage, Usability & Effect on Adherence and Clinical Outcomes of Text Message Reminders for Adolescents With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: CMSText (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20090445
Record Dates: First submitted 2010-11-29; First posted 2010-12-03 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison 1st (No Intervention): Not enrolled in the CMSText website text messaging system during last 3 months of study participation.
- Participant 1st (Experimental): Enrollment in the CMSText website text messaging system during first 3 months of study participation.
  Interventions: Other: Text Message Reminders

INTERVENTIONS:
Other: Text Message Reminders — During baseline (Participant 1st Arm) or Month 3 Visit (Comparison 1st Arm), the study staff member will demonstrate for the teen how to log-on to the calendar system and set up reminders. Teens will be able to set their own reminders and add other reminders in addition to those that are asthma related.
  Arms: Participant 1st

SUMMARY:
The purpose of this randomized crossover study is to determine the efficacy of participant designed medication reminders on asthma control, asthma related quality of life,and medication adherence. In addition, this study will provide data regarding the usage, usability, acceptability of an online system designed for creating text message reminders. It is hypothesized that the teens receiving text message reminders will report having greater quality of life related to their asthma, a reported increase in the control of their asthma, and increased adherence to their medication regimen compared to those teens that are not receiving the text message reminders.

DETAILED DESCRIPTION:
Adolescents are typically less adept at managing chronic illnesses and adhering to treatment plans than are parents of younger children. Adolescents are also typically "early adopters" to technological solutions and text messages are integral in today's teen culture. Text messages are gaining acceptance in health care both as appointment reminders and direct inquiries. The purpose of this randomized crossover study is to examine the effect of participant designed medication reminders on asthma control, asthma related quality of life, and medication adherence. In addition, this study will provide data regarding the usage, usability, and acceptability of an online system designed for creating text message reminders.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 12 and 22
* Diagnosis of Persistent Asthma
* Receiving care at Cincinnati Children's Hospital Medical Center or affiliate
* Prescription of a controller medication
* Must have a cell phone that receives text messages
* Asthma is not well-controlled based on ACT score
* English Speaking

Exclusion Criteria:

* No diagnosis of persistent asthma
* Receiving asthma care other than at a Cincinnati Children's Hospital Medical Center or affiliate
* Asthma is well-controlled based on ACT score
* Does not have a cell phone that receives text messages or plans to change phones within the next 6 months
* Is not taking a daily asthma controller medication
* Is currently receiving asthma appointment or medication reminder text messages from another source

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | Change from Baseline on ACT at 3 months (1st arm), Change from Baseline on ACT at 6 months (2nd arm)
  The teen will complete the Asthma Control Test (ACT), a validated 5-item Likert scale test that asks them to detail their asthma symptoms. These are questions consistent with those that would be asked by a clinician (i.e., how many times have you used your fast-acting inhaler in the past four weeks, how often does asthma limit your activities). The responses to these questions will also be used to calculate the teen's asthma control.

SECONDARY OUTCOMES:
The Pediatric Quality of Life Scale Version 4.0 Teen Report (ages 13- 18) (PedsQL) | Change from Baseline on PedsQL at 3 months (1st arm), Change from Baseline on PedsQL at 6 months (2nd arm)
  This assessment measures how much asthma has been a problem for them in the last month (i.e., "It is hard for me to be responsible for my medications.", "I worry about my asthma.")
Adherence | Change from Baseline in Adherence at 3 months (1st arm), Change from Baseline in Adherence at 6 months (2nd arm)
  Adherence to medication regimen will be monitored with the Smartinhaler Tracker developed by Nexus 6 ltd. It will record the adherence to medication administered through metered-dose inhalers, which include medication such as Qvar and Flovent. The Smartinhaler records the time and date medications were taken, whether the canister was shaken appropriately prior to inhalation, and how much the medication was inhaled.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Britto, M.D., M.P.H., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States